CLINICAL TRIAL: NCT02327507
Title: Bending the Oregon Health Plan (OHP) Dentistry Cost Curve in Central Oregon by Reducing the Burden of Oral Disease
Brief Title: Everybody Brush: A Community-wide Toothpaste Distribution Campaign
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Advantage Dental Services, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Advantage001
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Dental Caries
Keywords: children; fluoridated toothpaste; health education; Medicaid
MeSH Terms: conditions — Dental Caries; Health Education | interventions — Toothpastes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Toothpaste & Telephone Support: A tool kit with toothpaste and toothbrushes for the whole family along with oral hygiene instructions in both English and Spanish will be mailed to the homes of all OHP children and adolescents every three months. Half the populations will be assigned to also receive telephone support.
  Interventions: Behavioral: Toothpaste & Telephone Support
- Toothpaste only: A tool kit with toothpaste and toothbrushes for the whole family along with oral hygiene instructions will be mailed every three months

INTERVENTIONS:
Behavioral: Toothpaste & Telephone Support — Mailed toothpaste, messages and telephone support.
  Groups: Toothpaste & Telephone Support

SUMMARY:
Dental caries (tooth decay) is a disease with significant public health implications afflicting low-income children, with marked rural disparities in disease prevalence and treatment. More than 70% of 11th grade children in Crook, Deschutes and Jefferson counties have experienced tooth decay. Effective approaches to prevent decay include brushing with fluoridated toothpaste and professional dental care. Medicaid enrolled children are legally entitled to dental care under Early Periodic Screening, Diagnosis and Treatment (EPSDT), yet <50% had any care in 2010. Free distribution of toothpaste and toothbrushes combined with parental education can increase toothbrushing frequency and reducing tooth decay. However, many parents are confused about when to start, how much and often toothpaste should be used, and how to overcome behavioral difficulties in brushing toddlers' teeth or getting older children to brush their own. The investigators' objective is to implement and evaluate a community-wide toothpaste distribution campaign enhanced by telephone support for OHP children and adolescents and their families in Central Oregon

DETAILED DESCRIPTION:
A community-wide toothpaste distribution campaign enhanced by telephone support. A tooth kit with toothpaste and toothbrushes for the whole family together with oral hygiene instructions in English and Spanish will be mailed every 3 months. Half of the population will be randomly assigned to also receive telephone support (Short message service and one-to-one calls). Families will receive biweekly messages with oral hygiene tips. Bilingual culturally competent staff will be available by telephone to support families in overcoming barriers.

ELIGIBILITY:
Inclusion Criteria:

* Family speaks English or Spanish

Exclusion Criteria:

* None

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents enrolled in Medcaid OHP and assigned to Advantage Dental Services in Oregon in Crook, Deschutes, or Jefferson counties
Sampling Method: Non-Probability Sample
Enrollment: 21731 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
increased twice-a-day toothbrushing Toothbrushing | 1 year
  Parent reported toothbrushing frequency for child

SECONDARY OUTCOMES:
Satisfaction | 1 year
  Dental Satisfaction Questionnaire
Cost | 1 year
  Per member per month cost of care

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Milgrom, DDS, Principal Investigator — University of Washington
Locations (1):
- Advantage Dental Services, LLC, Redmond, Oregon, United States

REFERENCES:
- [Derived] Cunha-Cruz J, Milgrom P, Shirtcliff RM, Huebner CE, Ludwig S, Allen G, Scott J. "Everybody brush!": protocol for a parallel-group randomized controlled trial of a family-focused primary prevention program with distribution of oral hygiene products and education to increase frequency of toothbrushing. JMIR Res Protoc. 2015 May 22;4(2):e58. doi: 10.2196/resprot.4485. PMID 26002091